CLINICAL TRIAL: NCT00174265
Title: A Multicenter, Double-Blind, Flexible-Dose, 6-Month Extension Trial Comparing the Safety and Efficacy of Asenapine With Olanzapine in Subjects Who Completed Protocol A7501013
Brief Title: 6-Month Extension Trial of Asenapine With Olanzapine in Negative Symptoms Patients Who Completed the First 6- Month Trial (A7501014)(COMPLETED)(P05772)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05772; Aphrodite; A7501014
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asenapine (Experimental)
  Interventions: Drug: asenapine
- olanzapine (Active Comparator)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — 5-10 mg sublingually twice daily for 26 weeks
  Arms: asenapine
Drug: olanzapine — 5-20 mg by mouth once daily for 26 weeks
  Other Names: Zyprexa
  Arms: olanzapine

SUMMARY:
This is an extension study of A7501013 (P05771/NCT00145496) to further test

the efficacy and safety of Asenapine compared with a

marketed agent (olanzapine) in the treatment of patients with

persistent negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Continue to meet all demographic and procedural

inclusion criteria of the A7501013 trial to enter into

this extension trial.

* Have demonstrated an acceptable degree of compliance

and completed the A7501013 trial, and would benefit

from continued treatment according to the investigator.

Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant

medical condition.

* Have been judged to be medically noncompliant in the

management of their disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2005-07; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

REFERENCES:
- [Result] Buchanan RW, Panagides J, Zhao J, Phiri P, den Hollander W, Ha X, Kouassi A, Alphs L, Schooler N, Szegedi A, Cazorla P. Asenapine versus olanzapine in people with persistent negative symptoms of schizophrenia. J Clin Psychopharmacol. 2012 Feb;32(1):36-45. doi: 10.1097/JCP.0b013e31823f880a. PMID 22198451

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asenapine | Olanzapine
Started | 86 (85 participants received randomized treatment assignment and at least one dose of study medication.) | 110
Completed | 57 | 89
Not Completed | 29 | 21
Not completed — Adverse Event | 7 | 4
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other (Not specified) | 16 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine | Olanzapine | Total
Number analyzed (Participants) | 85 | 110 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 108 | 192
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 67 | 83 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Negative Symptoms of Schizophrenia Measured by the Negative Symptom Assessment (NSA) Scale Total Score
Description: The NSA Scale is a 16-item clinician-rated instrument for rating the negative symptomatology of schizophrenia. Total score ranges from 16 (best) to 96 (worst), with greater scores indicating greater severity of symptoms.
Time Frame: Baseline of A7501013 to Day 365
Population: Intent-to-treat (ITT) population. In-treatment change from baseline scores by visit and baseline scores from the ITT population are included in the Mixed Model for Repeated Measurements (MMRM) model.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 83 | 110
Units on a Scale
  Baseline | 61.5 (1.37) | 60.3 (1.20)
  Change from Baseline at Day 365 | -15.8 (1.48) | -11.0 (1.27)
Statistical Analysis 1: Comparison: Asenapine vs Olanzapine; The null hypothesis was that there was no difference in change from Baseline in NSA Scale total score between asenapine and olanzapine at Day 365; Test type: Superiority or Other; p = 0.0148, Mixed Model for Repeated Measurements — The test of hypothesis was a 2-tailed test with alpha=0.05 (0.049 to adjust for one interim analysis)

2. Secondary Outcome: Change From Baseline in Quality of Life Measured by the Quality of Life Scale (QLS) Total Score
Description: The QLS is a 21-item clinician-rated scale for rating psychosocial functioning (Interpersonal Relations, Instrumental Role, Intrapsychic Foundations, and Common Objects and Activities). The score ranges from 0 (worst) to 126 (best), with greater values indicating better quality of life.
Time Frame: Baseline of A7501013 to Day 365
Population: ITT population. In-treatment change from baseline scores by visit and baseline scores from the ITT population are included in the MMRM model.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 83 | 110
Units on a Scale
  Baseline | 45.3 (2.27) | 42.3 (1.99)
  Change from Baseline at Day 365 | 12.4 (2.05) | 11.7 (1.73)
Statistical Analysis 1: Comparison: Asenapine vs Olanzapine; The null hypothesis was that there was no difference in change from Baseline in QLS total score between asenapine and olanzapine at Week 52; Test type: Superiority or Other; p = 0.8100, Mixed Model for Repeated Measurements — Significant level adjusted for one interim analysis was set as 0.049 two-sided

ADVERSE EVENTS:
Arm/Group | Asenapine | Olanzapine
Serious Adverse Events (participants affected / at risk) | 4/85 | 4/110
Other Adverse Events (participants affected / at risk) | 14/85 | 31/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=85) | Olanzapine (N=110)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 3 (3)
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=85) | Olanzapine (N=110)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (10)
Weight Increased (Investigations) | 5 (5) | 13 (13)
Headache (Nervous system disorders) | 2 (2) | 8 (12)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for compelling legal reasons, neither the sponsor nor the investigator will communicate to third parties any result of the clinical trial before the clinical trial report has been released by the sponsor.